CLINICAL TRIAL: NCT00576095
Title: Hypothalamic-Pituitary-Adrenal (HPA)/ Dopamine Axis in Psychotic Depression
Brief Title: Clinical and Biological Characteristics of Psychotic Depression
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2R01MH050604-10 (NIH); MH50604; NCT00048269 (obsolete NCT alias); NCT00185926 (obsolete NCT alias)
Record Dates: First submitted 2007-12-14; First posted 2007-12-18 (Estimated); Last update posted 2014-03-14 (Estimated); Status verified 2014-03

CONDITIONS: Depression; Psychotic Disorders; Depressive Disorder, Major
MeSH Terms: conditions — Depression; Psychotic Disorders; Depressive Disorder, Major

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- PMD: Patients diagnosed with major depression with psychotic features
- NPMD: Patients diagnosed with major depression without psychotic features
- Controls: Participants with no psychiatric or depression history

SUMMARY:
The primary objective of this study is to investigate the relationships among findings in structural and functional neuroimaging, cognitive testing and HPA (hypothalamic-pituitary-adrenal) axis dysregulation in psychotic depression.

DETAILED DESCRIPTION:
Eligibility Procedures: Before entering the study and prior to any other procedures, you will be asked to read and sign this consent form. To determine if you are eligible for our study, you will then have a general medical (including menstrual cycle history on female patients) and psychiatric history taken, a physical examination your vital signs (blood pressure, pulse), height, weight, waist/hip ratio will be measured, and various psychiatric evaluations will be conducted. We will be video recording the psychiatric diagnostic assessment of every 5th patient who enrolls in our study.

On Day 1, your mood will be evaluated using a series of commonly used diagnostic instruments and rating scales. We will repeat the medical exam, blood and urine lab tests you had at your initial screening visit if it has been more than 4 weeks (30 days) since your eligibility screening.

The rest of the study includes an MRI, neuropsychological testing, questionnaires, and blood draws.

The MRI (called magnetic resonance imaging, MRI) involves having a picture of your brain taken using a magnet while a series of tasks is administered to you. The MRI scan procedures will take approximately 1 hour.

The neuropsychological testing consists of a series of tests to assess your memory and concentration (neuropsychological means the way your brain processes and completes specific tasks.) This testing, including directions, will take approximately 3 hours of your time. You will also be asked to complete several questionnaires during your hospital stay. These questionnaires ask for your views about your personality, your childhood experiences your quality of life, your mood and a variety of aspects of your daily functioning. The questionnaires may be completed anytime during your stay and will take about 2.5 hours to finish

The blood draws are done at the GCRC, where you will stay for 2 nights.

The following blood draw procedures will be performed for all participants on Day 1: At 4pm on Day 1, an intravenous line (IV; needle inserted into a vein) will be placed in your arm to draw hourly blood samples used for the measure of adrenocorticotropin (ACTH) and cortisol. ACTH is a hormone that controls the release of cortisol (a stress hormone) in your system and both of these hormones levels change under stressful conditions. The blood samples are taken in small amounts (approximately 1/2 teaspoon) and will be collected at 2pm and 4pm on Baseline Day 1, and then on the hour, every hour, starting at 6pm and ending at 9am the next day. A total of 72 ml(approximately 5 tablespoons) of blood will be drawn. The IV line will be removed following the last blood draw. If you presently live in a time zone different from the Pacific Standard Time zone (for example, Eastern Standard Time zone), we may begin taking hourly blood samples as early as 3pm on Baseline Day 1 in order to more accurately measure your body's daily rhythm of hormones.

The following blood draw procedures will be performed for all participants on Day 2: At 2pm on Baseline Day 2, you will have another IV line placed in your arm to draw hourly blood samples used for the measure of ACTH and Cortisol. At 3pm, you will be given 0.5mg (five 0.1mg tablets) of Fludrocortisone. Cortisol and ACTH are taken in small amounts (approximately 1/2 teaspoon) and will be collected on the hour, every hour, starting at 2 pm and ending at 7pm, then every 30 minutes until 12 midnight. Melatonin will be collected at 6:00pm, 7:00pm and then every 30 minutes until 12 midnight. Following the last blood draw, a blood sample will be taken for a clinical laboratory assessment to ensure your safety following Fludrocortisone administration. A total of 66ml's (4 1/2 tablespoons) of blood will be drawn. At 12 midnight, the IV line will then be removed and your vital signs will be taken.

ELIGIBILITY:
Inclusion Criteria:Inclusion criteria for PMD (individuals with Psychotic Major Depression) and NPMDs (individuals with Non-Psychotic Major Depression) are as follows:

1. DSM IV diagnosis of Major Depressive Disorder with or without psychotic features, Bipolar II Disorder with or without psychotic features in a major depressive episode.
2. 21-item HAM-D score greater than or equal to 21.
3. Thase Core Endogenomorphic Scale score greater than or equal to 6 on the items included in the 21-item HDRS.
4. Between 21 - 85 years of age.
5. If currently taking antipsychotic, antidepressant, anticonvulsant, and/or mood-stabilizing medications, must be stable on the medication for at least one-week prior to entering the study.
6. Pre-existing (current) primary treating psychiatrist for subjects with psychotic features.
7. Any secondary diagnoses from the anxiety disorder spectrum is acceptable. Primary pre-existing chronic Obsessive-Compulsive Disorder(OCD) will be an exclusion criteria.

Inclusion criteria for healthy controls are as follows:

1. Between 21 - 85 years of age. 2. Taking no medications 3. Have a HAM-D score of less than or equal to 5. Exclusion Criteria:Exclusion criteria for PMDs and NPMDs are as follows:

1. ECT in the 4 months prior to the study.
2. Abuse of drugs or alcohol in the 6 months prior to study.
3. Unstable or untreated hypertension, or cardiovascular disease.
4. If participating in the blood draw portion of the protocol, endocrine disorders are exclusionary.
5. Use of additional prescription medications, street drugs, or alcohol during the week before the study.
6. Any Axis II diagnosis or traits which would make participation in the study difficult.
7. Current pregnancy or lactation.

Exclusion criteria for healthy controls:

1. Personal history of Axis I or Axis II disorders.
2. Active unstable medical problems.
3. Abuse of drugs or alcohol in the 6 months prior to study.
4. Use of additional prescription medications, street drugs, or alcohol during the week before the study.
5. Currently pregnant or lactating.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Major depression with psychosis Major depression without psychosis Healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2005-08; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Cortisol | baseline
  Hourly serum cortisol

SECONDARY OUTCOMES:
Cognitive function | Baseline
  Standard domains - including verbal memory, executive functioning, attention

CONTACTS AND LOCATIONS:
Overall Officials: Alan Schatzberg, Principal Investigator — Stanford University; Jennifer Keller, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Derived] Cherian K, Schatzberg AF, Keller J. HPA axis in psychotic major depression and schizophrenia spectrum disorders: Cortisol, clinical symptomatology, and cognition. Schizophr Res. 2019 Nov;213:72-79. doi: 10.1016/j.schres.2019.07.003. Epub 2019 Jul 12. PMID 31307859
- [Derived] Keller J, Gomez R, Williams G, Lembke A, Lazzeroni L, Murphy GM Jr, Schatzberg AF. HPA axis in major depression: cortisol, clinical symptomatology and genetic variation predict cognition. Mol Psychiatry. 2017 Apr;22(4):527-536. doi: 10.1038/mp.2016.120. Epub 2016 Aug 16. PMID 27528460